CLINICAL TRIAL: NCT04838132
Title: Application of Transversus Thoracis Muscle Plane Block Plus Rectus Sheath Block in the Perioperative Pain Management of Cardiac Surgery : Study Protocol of a Randomized Double-blind Controlled Trial
Brief Title: Transversus Thoracis Muscle Plane Block Plus Rectus Sheath Block in the Perioperative Pain Management of Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-2021-009-01
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Bypass Grafting or Heart Valve Surgery Via Median Sternotomy
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transversus thoracis muscle plane and rectus sheath block with ropivacaine (Experimental): Using the plane technique to place a 22-gauge, 80-mm needle obliquely upwards until the needle tip is located at the plane between the internal intercostal muscles and the transverse pectoralis muscle (TTP block) and rectus sheath block, give 15ml and 10ml 0.3% ropivacaine respectively.
  Interventions: Procedure: Bilateral transversus thoracis muscle plane and rectus sheath block with ropivacaine
- Transversus thoracis muscle plane and rectus sheath puncture with saline (Experimental): Using the plane technique to place a 22-gauge, 80-mm needle obliquely upwards until the needle tip is located at the plane between the internal intercostal muscles and the transverse pectoralis muscle (TTP block) and rectus sheath block, give 15ml and 10ml 0.9% saline respectively.
  Interventions: Procedure: Bilateral transversus thoracis muscle plane and rectus sheath puncture with saline

INTERVENTIONS:
Procedure: Bilateral transversus thoracis muscle plane and rectus sheath block with ropivacaine — A linear array transducer (6-13 MHz) with a sterile cover and a 22-gauge (G) block needle (KDL™, Kindly group, Shanghai, China) will be used. Place the ultrasound probe on the longitudinal plane 1 cm outside the edge of the sternum in the fourth intercostal space, and identify the T3-T4 intercostal space under ultrasound. Use the plane technique to place a 22-gauge, 80-mm needle obliquely upwards until the needle tip is located at the plane between the internal intercostal muscles and the transverse pectoralis muscle. After general anesthesia, all subjects were injected with 0.3% ropivacaine 15ml and 10ml respectively after insertion of a needle into bilateral transverse thoracic muscle plane and rectus sheath guided by B-ultrasound.
  Arms: Transversus thoracis muscle plane and rectus sheath block with ropivacaine
Procedure: Bilateral transversus thoracis muscle plane and rectus sheath puncture with saline — A linear array transducer (6-13 MHz) with a sterile cover and a 22-gauge (G) block needle (KDL™, Kindly group, Shanghai, China) will be used. Place the ultrasound probe on the longitudinal plane 1 cm outside the edge of the sternum in the fourth intercostal space, and identify the T3-T4 intercostal space under ultrasound. Use the plane technique to place a 22-gauge, 80-mm needle obliquely upwards until the needle tip is located at the plane between the internal intercostal muscles and the transverse pectoralis muscle. After general anesthesia, all subjects were injected with 0.9% saline 15ml and 10ml respectively after insertion of a needle into bilateral transverse thoracic muscle plane and rectus sheath guided by B-ultrasound.
  Arms: Transversus thoracis muscle plane and rectus sheath puncture with saline

SUMMARY:
An emerging regional block technique, transverse thoracic muscle block covers the T2-T6 intercostal nerves and can effectively relieve perioperative pain during median sternotomy. Bilateral transverse thoracic muscle plane( TTP) block is expected to be a new analgesic mode in perioperative of cardiac surgery via sternotomy.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, parallel controlled clinical trial. Eighty patients planning to undergo coronary artery bypass grafting or heart valve surgery via median sternotomy were randomly assigned 1:1 to the experimental group or control group. After general anesthesia, all subjects were injected with 0.3% ropivacaine (experimental group) or 0.9% normal saline (control group) 15ml and 10ml respectively after insertion of a needle into bilateral transverse thoracic muscle plane and rectus sheath guided by B-ultrasound by anesthesiologist. The main outcome indicators were the threshold of incision pain and the total amount of analgesics used during the operation and 48h after the operation. Secondary outcome measures were as follows: postoperative VAS score, duration of mechanical ventilation, days in ICU, total days of hospitalization, and hospitalization cost. This study will provide evidence-based medical evidence and clinical data support for the application of TTP block in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily cooperate with the study and sign an informed consent form;
* Ages between 18 and 65;
* American Society of Anesthesiologists (ASA) classification: I-III;
* Undergo coronary artery bypass grafting (CABG) or heart valve surgery with midsternal incision.

Exclusion Criteria:

* Refuse to participate in the trial;
* Allergic to the anesthetics or analgesics;
* Suffering with serious systemic diseases (kidney, liver, lungs and endocrine system);
* American Association of Anesthesiologists (ASA) classification: IV-V;
* Unstable hemodynamics;
* History of drug abuse or chronic pain;
* Mental disorders or communication difficulties;
* Died during or immediately after the operation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hyperalgesia | Surgery to 48 hours after
  a 180mN von-Frey wire (Touch Test™ Sensory Evaluator, USA) was used to test the pain sensitivity of the area around the wound
The total amount of analgesics used in the perioperative period. | Surgery to 48 hours after
  During the perioperation, the amount of analgesics during the operation, the total amount of analgesic pump drugs used and the frequency of pressing the additional bolus trigger in the patient's analgesia system at 48 hours after the operation, and the amount of remedial analgesics

SECONDARY OUTCOMES:
Visual Analogue Scale | Extubation to 24 hours after
  A scale with a length of about 10cm is used. One side is marked with 10 scales, and the two ends are marked with "0" and "10" points respectively. 0 points mean painless, and 10 points mean the most intense pain that is unbearable
Length of stay in hospital | the day before hospital discharge
  record how many days doses the patient spends in hospital
Postoperative complications | the day before hospital discharge
  such as nausea and vomiting, pulmonary infection, wound infection, delayed healing, renal insufficiency, etc.
incidence of postoperative delirium | Day 7 after operation
  Changes in postoperative state of consciousness were assessed

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zheng, doctor, Study Chair — Guangzhou First People's Hospital
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China